**IRAS ID:** 



320293



## **Participant Informed Consent Form**

| Trial Name:<br>Chief<br>Investigator:<br>Principal | Evaluation of Pilot Online Binge Eating Disorder Group in under 18s. Dominique Muhumuza Dominique Muhumuza | | | | | |
|---|---|---|---|---|---|---|
| | | | | | Investigator: Participant Ide | · |
| | | | | | number: | |
| | | | | Please<br>initial<br>each box | | |
| 1. I confirm th | nat I have: | | | | | |
| | nderstand the information sheet <b>PIS</b> and for the above study. | Service User | - BE Group Intervention | | | |
| <ul> <li>had enough<br/>think are re</li> </ul> | h time to think whether or not I want teasonable. | o take part, as | sk questions and get answers that I | | | |
| have been | I that this study is designed to further<br>approved by the Research Ethics Co<br>nmittee of Coventry Warwickshire Par | mmittee of Ne | ewman University and Research | | | |
| I understand that my taking part is voluntary and that I am free to stop taking part at any time without giving any reason, without my medical care or legal rights being affected. | | | | | | |
| | try and complete the questionnaires. | I understand | that I can take a break or stop | | | |
| 4. I understar | nd that: | | | | | |
| I am partici | ipating in a group | | | | | |
| I will be asl | ked to complete weekly tasks as part | of the group i | ntervention | | | |
| • I do not wa | int my parents to be involved in this re | esearch projed | et. | | | |
| I understand that my questionnaires and feedback may be looked at by people from the Coventry and Warwickshire Partnership trust or Newman University. I give permission for these individuals to have access to all information collected. | | | | | | |
| 6. I do not ag | o not agree to my parents/carer being contacted about this study. | | | | | |
| something | rstand that information collected will be kept confidential. However, if I tell the researchers hing they think is likely to result in immediate harm to myself or others, they may have to me about disclosing this in line with the law and local safeguarding procedures. | | | | | |
| 8. I agree the | 8. I agree the ED team to inform my GP that I am participating in this project. | | | | | |
| 9. I agree to | take part in the above study. | | | | | |
| Your name (in | capitals) | Date | Signature | | | |
| Name of persor | n taking consent (in capitals) | Date | Signature | | | |
| Name of persor | n recording consent (if different) | Date | Signature | | | |
| (III Capitals) | | | | | | |

When completed, the original should be kept in the Investigator Site File, a copy should be given to the patient and one kept in the study notes along with the Participant Information Sheet.